CLINICAL TRIAL: NCT05547347
Title: A Phase 1 Study in Patients With Clinically Node-Positive Breast Cancer to Assess the Safety, Ultrasound Conspicuity, and Migration of an Ultrasound Twinkling Marker Obeservedfor Sonographic Targeting (UTMOST TRIAL)
Brief Title: Safety, Ultrasound Conspicuity, and Migration of Twinkling Markers in Patients With Locally Advanced Breast Cancer
Status: Suspended | Type: Observational
Why Stopped: Pending biocompatibility testing
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-002857; NCI-2022-06278 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); DTP (Other: Mayo Clinic Radiology)
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Locally Advanced Breast Carcinoma; Resectable Breast Carcinoma
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Observational (twinkle marker placement): Patients undergo percutaneous ultrasound-guided breast clip placement with a conventional biopsy marker (if not already present) and a twinkling marker throughout the trial. Patients undergo a breast ultrasound during screening, on study, and as clinically indicated. Patient also undergoes a mammogram on study and as clinically indicated as well as a MRI as clinically indicated.
  Interventions: Procedure: Magnetic Resonance Imaging; Procedure: Mammogram; Procedure: Ultrasound; Procedure: Ultrasound-Guided Biopsy; Device: Twinkle marker

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Mammogram — Undergo a mammogram
Procedure: Ultrasound — Undergo a breast ultrasound
Procedure: Ultrasound-Guided Biopsy — Undergo a percutaneous ultrasound-guided breast clip placement
  Other Names: Ultrasound Guided Biopsy
Device: Twinkle marker — Patients undergo percutaneous ultrasound-guided breast clip placement with a conventional biopsy marker (if not already present) and a twinkling marker on study.

SUMMARY:
This phase I study assesses the safety, ultrasound visibility (conspicuity), and movement from normal position (migration) of the twinkling marker in patients with breast cancer that has spread to the axillary lymph nodes (locally advanced) who will be undergoing neoadjuvant systemic therapy and surgery. Biopsy markers are used to identify the sites of cancer involvement in both the breasts and lymph nodes. These biopsy markers are needed to help guide breast cancer surgery. Twinkling markers are designed to have the same size and shape of conventional biopsy markers, but are made of a radio-opaque material that assists with localization of the marker. The twinkling marker may make it more easily seen with ultrasound at the time of breast cancer surgery as compared to conventional biopsy markers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To show that the biologically inert, Food and Drug Administration (FDA)-approved material that comprises the Mayo-developed twinkling marker, either pre-made and sterilized or made immediately before placement, (Patent Application Title: Non-Metallic Ultrasound-Detectable Markers Patent Application No.: 62/903,078, Application Type: Provisional) remains conspicuous under ultrasound after neoadjuvant systemic therapy in patients with clinically node-positive breast cancer.

SECONDARY OBJECTIVE:

I. To evaluate the safety and migration of the Mayo-designed twinkling marker in patients during neoadjuvant systemic therapy (NST).

OUTLINE:

Patients undergo percutaneous ultrasound-guided breast clip placement with a conventional biopsy marker (if not already present) and a twinkling marker throughout the trial. Patients undergo a breast ultrasound during screening, on study, and as clinically indicated. Patient also undergoes a mammogram on study and as clinically indicated as well as a magnetic resonance imaging (MRI) as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years or older with breast cancer and biopsy-proven malignant involvement of an axillary lymph node
* Surgical management will be determined by the surgeon, who will decide if preoperative I-125 seed localization of the positive node is necessary or if they will retrieve the positive node with intraoperative ultrasound guidance. During surgery, the targeted node, its associated biopsy markers, I-125 seed if placed, and twinkling marker will be resected. The position of the marker in the lymph node or proximity to the node will be noted from the surgical and pathology documentation.
* Surgery will be performed by one of the surgeons in the Division of Breast and Melanoma Surgical Oncology (Dr. Judy Boughey, Dr. Amy Degnim, Dr. Tina Hieken, Dr. Jeffrey Johnson, Dr. Mary Mrdutt, Dr. Dalliah Black, Dr. Mara Piltin)
* Patients must be able to understand the study procedures and comply with them for the entire length of the study
* No contraception is necessary or required

Exclusion Criteria:

* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent
* Current or past participation within a specified timeframe in another clinical trial, as warranted by the administration of this intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced breast cancer patients undergoing neoadjuvant systemic therapy and surgery with Dr. Piltin at Mayo Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Long-term efficacy of the twinkling marker | through study completion, an average of 4 months
  The primary outcome is information on the long-term efficacy of the twinkling marker in humans placed in the lymph nodes of patients undergoing neoadjuvant systemic therapy (NST) for breast cancer. The data will explore the presence/absence of the twinkling artifact associated with the twinkling marker under ultrasound.

SECONDARY OUTCOMES:
Determination of safety and migration of the twinkling marker | through study completion, an average of 4 months
  The secondary outcome is determination of safety and migration of the Mayo-designed twinkling marker in patients after NST. Clinical notes will be reviewed to assess for any complications related to the twinkling marker during NST. Migration will be determined from surgical and pathology documentation.

CONTACTS AND LOCATIONS:
Overall Officials: Christine U Lee, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials